CLINICAL TRIAL: NCT05238571
Title: Somatosensory Outcomes Following Re-surgery in Persistent Severe Pain After Groin Hernia Repair
Brief Title: Does Re-surgery Improve Somatosensory Outcomes in Persistent Pain After Groin Hernia Repair
Status: Completed | Type: Observational
Sponsor: mads u werner (Other)
Responsible Party: Sponsor-Investigator, mads u werner, Principal Investigator, MD, DMSci, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: H-2-2011-023-FE
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Patients With Persistent Severe Pain After Groin Hernia Repair
Keywords: groin hernia repair; chronic post-surgical pain; pain thresholds; patient reported outcome measures; reoperation; sensory thresholds
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Re-surgery — Re-surgery with meshectomy and selective neurectomy

SUMMARY:
Groin hernia repair is accompanied by persistent severe pain in 2-4% of the patients significantly restraining psychophysical functions. Re-surgery with meshectomy and selective neurectomy may improve the pain condition, compared to non-surgical alternatives. In the current study, the primary objective was to examine and describe the underlying pathophysiological perturbations by quantitative somatosensory testing before and after re-surgery.

DETAILED DESCRIPTION:
Persistent severe pain occurring in the aftermath of a surgical procedure is frequently associated with significant impairment of physical and psycho-social functions. After groin hernia repair (GHR), 2-4% of patients develop persistent severe pain. The GHR procedure, previously considered belonging to "minor" surgeries, qualifies as a rather complex procedure performed in a territory with a high density of nerve fibers, accommodating essential functions for locomotion and reproduction. More than 20 million repairs are performed annually worldwide, and consequently, it is estimated that 400.000-800.000 patients each year will develop persistent severe pain after the groin hernia repair (PSPG). Management of PSPG is medically challenging and may require re-surgery with mesh removal and selective neurectomy. After re-surgery for pain after open primary GHR, a potential pain-relieving effect, as well as an improvement of the deteriorated physical functions, has been demonstrated.

Quantitative somatosensory testing (QST) is an investigational psychophysiological tool with the potential to uncover the putative pathophysiological substrate in PSPG, i.e., neuropathic and inflammatory constituents. The method may also be used to quantitate changes induced by the re-surgery. Since re-surgery is a neuroablative procedure, essentially performed in previously damaged tissue, it is of interest to examine the extent of neurological perturbations, i.e., 'loss' and 'gain' of sensory functions and the relation to clinical outcome measures.

The authors are only aware of one previous PSPG-study (n = 21) finding that re-surgery, including meshectomy and selective neurectomy, was associated with increased pain pressure thresholds, decreased pain ratings and improved pain-related functional measures. The objectives of the current study, comparing pre with post-re-surgery data, were first to perform a more detailed analysis of the quantitative somatosensory data regarding 'loss' and 'gain' of sensory functions and their relation to clinical outcome measures. Second, to corroborate the clinical outcome findings of the previous study using a threefold larger cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent severe pain (activity-related or maximal pain intensity > 7 NRS-scores [numeric pain rating scale 0-10]) following unilateral, uncomplicated, open groin hernia repair.

Exclusion Criteria:

* All that contradicts the above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent severe pain after groin hernia repair.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-04-24 (Actual); Primary Completion 2015-03-19 (Actual); Study Completion 2015-03-19 (Actual)

PRIMARY OUTCOMES:
Thermal thresholds | 3-6 months
  Warmth detection threshold (WDT), cool detection threshold, heat pain threshold (HPT) and cold pain threshold (CPT) are made by a computerized contact thermode (Thermotest, Somedic AB, Sweden) with an active thermal surface of 12.5 cm^2 (2.5 x 5.0 cm^2). The thresholds are determined from a baseline temperature of 32°C with a ramp rate of + 1°C/s. Cut-offs for heat and cold are 50°C and 5°C, respectively. The assessments are made in triplicate and the mean values are used in the statistical analyses.
Pressure algometry | 3-6 months
  Deep-tissue pain sensitivity is assessed using a hand-held pressure algometer with a neoprene-coated tip of area 1.0 cm2 (Somedic AB, Sweden), as previously described. The algometer is applied perpendicularly to the skin with a pressure rate of 30 kPa/s. The study subject is told to report the pressure pain threshold (PPT) by activating the button device when pain is perceived. The cut-off limit is 350 kPa. Testing is done in triplicate and the average value is used in the statistical analyses.
Suprathreshold heat stimulation | 3-6 months
  A short tonic heat stimulus (heating area 12.5 cm^2; ramp rate: 1°C/s, plateau: 47°C, 5 s; STH) is delivered in order to evaluate the suprathreshold heat pain perception (NRS).
Temporal summation | 3-6 months
  Temporal summation test, i.e., the perception in response to repetitive (0.3 to 3 Hz) mechanical stimulation [i.e., wind-up like pain: WUP], indicates presence of central sensitization. The repetitive 1 Hz stimuli for 60 s are either dynamically delivered by a brush or statically delivered by a polyamide filament (one nominal rank below TPT). The study subjects are told to report the level of pain (NRS) every 15 s-1 during the stimulation. Signs of aftersensations are followed 60 s after discontinuation of the stimulation, and the intensity of discomfort or pain is rated by NRS.

SECONDARY OUTCOMES:
Activity Assessment Scale (AAS) | 3-6 months
  Changes in AAS scores before and thre-six months after operation
Pain intensity scores (NRS) | 3-6 months
  Changes in pain intensity scores (NRS) at rest, on average and maximally before and thre-six months after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Multidisciplinary Pain Center, Neuroscience Center, Copenhagen University Hospital, DENMARK, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available as a supplement to the published scientific article.

REFERENCES:
- [Background] Bande D, Molto L, Pereira JA, Montes A. Chronic pain after groin hernia repair: pain characteristics and impact on quality of life. BMC Surg. 2020 Jul 6;20(1):147. doi: 10.1186/s12893-020-00805-9. PMID 32631293
- [Background] Chapman CR, Vierck CJ. The Transition of Acute Postoperative Pain to Chronic Pain: An Integrative Overview of Research on Mechanisms. J Pain. 2017 Apr;18(4):359.e1-359.e38. doi: 10.1016/j.jpain.2016.11.004. Epub 2016 Nov 28. PMID 27908839
- [Background] Campanelli G, Bruni PG, Morlacchi A, Cavalli M. Chronic Pain after Inguinal Hernia Repair. In: Campanelli G, editor. Inguinal Hernia Surgery. Milano: Springer Milan; 2017. p. 157-68.
- [Background] Nikkolo C, Kirsimagi U, Vaasna T, Murruste M, Suumann J, Seepter H, Lepner U. Prospective study evaluating the impact of severity of chronic pain on quality of life after inguinal hernioplasty. Hernia. 2017 Apr;21(2):199-205. doi: 10.1007/s10029-016-1569-4. Epub 2016 Dec 26. PMID 28025741
- [Background] HerniaSurge Group. International guidelines for groin hernia management. Hernia. 2018 Feb;22(1):1-165. doi: 10.1007/s10029-017-1668-x. Epub 2018 Jan 12. PMID 29330835
- [Background] Jorgensen SG, Oberg S, Rosenberg J. Treatment of longstanding groin pain: a systematic review. Hernia. 2019 Dec;23(6):1035-1044. doi: 10.1007/s10029-019-01919-7. Epub 2019 Feb 28. PMID 30820781
- [Background] Andresen K, Rosenberg J. Management of chronic pain after hernia repair. J Pain Res. 2018 Apr 5;11:675-681. doi: 10.2147/JPR.S127820. eCollection 2018. PMID 29670394
- [Background] Jensen EK, Ringsted TK, Bischoff JM, Petersen MA, Rosenberg J, Kehlet H, Werner MU. A national center for persistent severe pain after groin hernia repair: Five-year prospective data. Medicine (Baltimore). 2019 Aug;98(33):e16600. doi: 10.1097/MD.0000000000016600. PMID 31415351
- [Background] Werner MU. Management of persistent postsurgical inguinal pain. Langenbecks Arch Surg. 2014 Jun;399(5):559-69. doi: 10.1007/s00423-014-1211-9. Epub 2014 May 23. PMID 24849039
- [Background] Bischoff JM, Enghuus C, Werner MU, Kehlet H. Long-term follow-up after mesh removal and selective neurectomy for persistent inguinal postherniorrhaphy pain. Hernia. 2013 Jun;17(3):339-45. doi: 10.1007/s10029-013-1073-z. Epub 2013 Mar 15. PMID 23494661
- [Background] Aasvang E, Kehlet H. Surgical management of chronic pain after inguinal hernia repair. Br J Surg. 2005 Jul;92(7):795-801. doi: 10.1002/bjs.5103. PMID 15962258
- [Background] Aasvang EK, Kehlet H. The effect of mesh removal and selective neurectomy on persistent postherniotomy pain. Ann Surg. 2009 Feb;249(2):327-34. doi: 10.1097/SLA.0b013e31818eec49. PMID 19212190
- [Background] Linderoth G, Kehlet H, Aasvang EK, Werner MU. Neurophysiological characterization of persistent pain after laparoscopic inguinal hernia repair. Hernia. 2011 Oct;15(5):521-9. doi: 10.1007/s10029-011-0815-z. Epub 2011 Apr 9. PMID 21479588